CLINICAL TRIAL: NCT01072383
Title: A Randomized, Placebo-controlled, Double-blind, Multicentre, Multiple Dose, Cohort Study With Escalating Doses to Evaluate the Safety and Efficacy of the Humanized Monoclonal Antibody BT061 Administered to Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: Safety and Efficacy of Multiple Doses of BT061 in Patients With Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biotest (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 973
Record Dates: First submitted 2010-02-18; First posted 2010-02-22 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Psoriasis Vulgaris
Keywords: chronic plaque psoriasis; psoriasis vulgaris; autoimmune disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BT061 (Experimental): receiving BT061 (active compound)
  Interventions: Drug: BT061
- Placebo (Placebo Comparator): receiving a placebo
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: BT061 — administration of BT061 either intravenous or subcutaneous
  Other Names: SC or IV administration of BT061 or placebo
  Arms: BT061
Drug: placebo treatment — administration of the end formulation buffer of BT061 without active ingredient, either subcutaneous or intravenous
  Other Names: SC or IV administration of BT061 or placebo
  Arms: Placebo

SUMMARY:
This Phase II clinical study is to test safety and efficacy of BT061 against psoriasis given as repeated doses.

DETAILED DESCRIPTION:
Patients are enrolled into escalating dose levels. Improvement of PASI, physician's global assessment and itching score is evaluated after administration of BT061 or placebo. Safety data are assessed by an independent data and safety monitoring board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with moderate, moderate to severe or severe chronic plaque psoriasis diagnosed ≥ 12 months prior to Screening.
* BSA (Body surface area) involvement > 10% for more than 6 months.
* PASI ≥10.
* Age ≥ 18 to ≤ 75 years.
* Body mass index (BMI) of 18-30 kg/m2 with a body weight between 50 and 130 kg.

Exclusion Criteria:

* Erythrodermic, guttate or palmar pustular psoriasis (mixed forms may be admissible if chronic plaque psoriasis clearly remains the predominant diagnosis
* Treatment with a biological within less than 30 days or within less than 5 half-lives of the respective compound prior to administration of BT061/placebo.
* Serious local (e.g. abscess) or systemic infection (e.g. pneumonia, septicaemia) within 3 months prior to the administration of BT061 or placebo.
* Presence or history of clinically significant immune deficiency or autoimmune disease (except psoriasis).
* Positive diagnosis for acute or chronic infections (i.e. Hepatitis C Virus [HCV], Hepatitis B Virus [HBV], Human Immunodeficiency Virus [HIV]) at Screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-02; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Improvement in PASI score (Psoriasis Area and Severity Index) , as compared to PASI at baseline visit, | weekly during treatment, then 1 week, 1 month and 3 months after last dosing

SECONDARY OUTCOMES:
Dose group with the highest number of responders (PASI score improvement) | weekly during treatment, then 1 week, 1 month and 3 months after last dosing
PGA (Physician's global assessment) | weekly during treatment, then 1 week, 1 month and 3 months after last dosing
Itching score | weekly during treatment, then 1 week, 1 month and 3 months after last dosing
DLQI (dermatology life quality index) | weekly during treatment, then 1 week, 1 month and 3 months after last dosing
Physical examination | weekly during treatment, then 1 week, 1 month and 3 months after last dosing
Differential white blood cell count | weekly during treatment, then 1 week, 1 month and 3 months after last dosing
Cytokine profile | weekly during treatment, then 1 week after last dosing

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Kemény, M.D., Principal Investigator — Szegedi Tudományegyetem (Study site)
Locations (13):
- Czechia (5):
  - Dermatologic Clinic, Ostrava
  - Dermatologic Clinic I, Prague
  - Dermatologic Clinic Prague III, Prague
  - Dermatologic Clinic Prague II, Prague
  - Dermatologic Clinic, Ústí nad Labem
- Hungary (8):
  - Dermatologic Clinic, Budapest
  - Dermatologic Clinic, Debrecen
  - Dermatologic Clinic, Miskolc
  - Dermatologic Clinic, Szeged
  - Dermatologic Clinic, Szikszó
  - Dermatologic Clinic, Szolnok
  - Dermatologic Clinic, Szombathely
  - Dermatologic Clinic, Veszprém